CLINICAL TRIAL: NCT02759367
Title: Adequate Intake of Potassium Does Not Cause Hyperkalemia in Hypertensive Individuals on Medications That Antagonize the Renin Angiotensin Aldosterone System
Brief Title: Increasing Potassium Intake in Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSH 08-0025-A
Record Dates: First submitted 2015-12-22; First posted 2016-05-03 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Nutrition; Potassium
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Masking Description: Treating physicians and participants were not blinded to randomization. Investigators performing randomization and analysis of dietary intake were blinded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High potassium diet group (Experimental): Individuals in this arm were asked to increase dietary potassium intake over a 4 week period. This was achieved through an increase in consumption of fruits and vegetables.
  Interventions: Other: High potassium diet
- Usual diet group (No Intervention): Individuals in this group were asked to continue habitual dietary intake.

INTERVENTIONS:
Other: High potassium diet — An increase in consumption of high potassium fruits and vegetables
  Arms: High potassium diet group

SUMMARY:
This study evaluates the safety of increasing dietary potassium intake in a hypertensive population that may be at risk for hyperkalemia.

DETAILED DESCRIPTION:
The blood pressure lowering benefits of increasing dietary potassium (K⁺) are well known. As such dietary recommendations for hypertension focus on a diet rich in high K⁺ food sources such as fruits and vegetables. An important theme to be addressed is the safety of achieving high dietary K⁺ intake in hypertensive individuals who are also receiving medical therapy that might predispose to elevated serum K⁺ levels (hyperkalemia).

The purpose of this study was to assess the impact of aggressively increasing dietary K⁺ on serum K⁺ concentrations in hypertensive individuals with intact renal function medicated with RAAS blocking drugs. The investigators hypothesized that dietary K⁺ supplementation would not provoke hyperkalemia despite treatment with either an angiotensin converting enzyme (ACEi) or an angiotensin receptor blocker (ARB).

The investigators conducted an open controlled clinical trial in 20 hypertensive subjects with normal renal function who were randomized to a usual diet group (UD n=10), or a high potassium diet group (HKD, n= 10). Fruits and vegetables were used to increase potassium intake. All participants were on an ACEi or and ARB. Serum potassium concentration, 3- day food records and 24 Hour urine collections were completed at baseline and at the end of the 4-week study.

ELIGIBILITY:
Inclusion Criteria:

* Medically treated hypertension as diagnosed Hypertension was established by the participant's cardiologist or if recruited from the online community hypertension was self-reported and confirmed by study investigators based on participant's medical prescription.
* Treatment with an beta blocker, ACE inhibitor, or angiotensin receptor blocker without any adjustment over the previous 3 months
* K+ intake at baseline of less than 80 mmol/day (food diary of 24 hour food recall).

Exclusion Criteria:

* Patients with an episode of acute coronary syndrome, or revascularization within the previous 3 months will not be included.
* Serum K+ concentration 5.0 mmol/L
* Serum creatinine > 130 mmol/L.
* Inability to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Serum potassium concentration | 4 weeks

SECONDARY OUTCOMES:
24 hour urinary potassium excretion | 4 weeks
3 day dietary food diary | 4 weeks
  Food record will assess marco and mirco nutrient intake.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malta D, Arcand J, Ravindran A, Floras V, Allard JP, Newton GE. Adequate intake of potassium does not cause hyperkalemia in hypertensive individuals taking medications that antagonize the renin angiotensin aldosterone system. Am J Clin Nutr. 2016 Oct;104(4):990-994. doi: 10.3945/ajcn.115.129635. Epub 2016 Aug 31. PMID 27581475